CLINICAL TRIAL: NCT06066372
Title: Application of Machine Learning Models to Reduce Need for Diagnostic EUS or MRCP in Patients With Intermediate Likelihood of Choledocholithiasis- A Prospective, Open Label, Diagnostic Study
Brief Title: Application of Machine Learning Models to Reduce Need for Diagnostic EUS or MRCP in Patients With Intermediate Likelihood of Choledocholithiasis
Status: Recruiting | Type: Observational
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Other Study IDs: AI EUS Choledocholithiasis
Record Dates: First submitted 2023-09-13; First posted 2023-10-04 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Choledocholithiasis
MeSH Terms: conditions — Choledocholithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Machine learning predictive model can help in stratifying heterogenous intermediate likelihood group to reduce need for EUS or MRCP in selected subgroup of patients.

DETAILED DESCRIPTION:
The current guidelines for suspected choledocholithiasis are aimed to reduce the risk of patient receiving diagnostic ERCP and reduce the risk of post ERCP adverse events. In this process there is apparent increase in number of patients in the intermediate likelihood group requiring EUS or MRCP. This can increase the health care utilization and cost of care for intermediate likelihood patients. The field of artificial intelligence in clinical medicine is evolving rapidly. The use of artificial intelligence based machine learning model is not adequately studied for prediction of choledocholithiasis. Machine learning predictive model can help in stratifying heterogenous intermediate likelihood group to reduce need for EUS or MRCP in selected subgroup of patients.

ELIGIBILITY:
Inclusion Criteria:

• Individual 18 years or older with a suspected choledocholithiasis satisfying either ASGE or ESGE risk stratification criteria of intermediate likelihood undergoing EUS or MRCP

Exclusion Criteria:

* Patients having co-exiting disease of pancreato biliary system other than gall stones and choledocholithiasis which include chronic pancreatitis, biliary stricture, pancreatobiliary malignancy, portal biliopathy
* Patients having underlying chronic liver diseases
* Pregnancy and breast feeding
* Previous history of cholecystectomy

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with suspected choledocholithiasis satisfying either ESGE or ASGE risk stratification criteria of intermediate likelihood of choledocholithiasis will be prospectively enrolled from AIG Hospitals, Hyderabad
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Area Under the Receiver Operating Characteristic Curve (AUROC) of the Machine Learning Model | 1 month
  Area under the receiver operating characteristic curve (AUROC) of the machine learning-based prediction model for identifying the presence of choledocholithiasis.

SECONDARY OUTCOMES:
Diagnostic Accuracy Metrics of Endoscopic Ultrasound (EUS) or Magnetic Resonance Cholangiopancreatography (MRCP) | 1 Month
  Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and area under the receiver operating characteristic curve (AUROC) of magnetic resonance cholangiopancreatography (MRCP) for identification of choledocholithiasis.
Validation Performance of the Machine Learning Prediction Model | 1 Month
  Validation performance of the machine learning model for predicting choledocholithiasis, assessed using AUROC, calibration metrics (Brier score), and calibration plots in an independent validation cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Mohan Ramchandani, MD, Study Director — Asian Institute of Gastroenterology
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, Telangana, India